CLINICAL TRIAL: NCT05281445
Title: Exploring the Role of Neuroactive Steroids in Tourette Syndrome
Acronym: NS in TS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Utah (Other)
Collaborators: University of Miami (Other); Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Marco Bortolato, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00150143
Record Dates: First submitted 2022-02-24; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Tourette Syndrome in Children

STUDY DESIGN:
Intervention Model Description: Tic suppression task
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tic suppression (Experimental): Children with tics will undergo a tic suppression experimental paradigm.
  Interventions: Behavioral: Tic suppression task

INTERVENTIONS:
Behavioral: Tic suppression task — Tic Suppression Task (TST, administered to Tourette syndrome participants only): At the beginning of the task, the child participant will be seated alone in front of a computer monitor with a countdown timer visible on the screen. For the first 10 minutes (baseline condition) they will be asked to tic freely and not to try to suppress their tics. For the second 10 minutes children will be asked to suppress their tics and will receive points for successful suppression. Participants will then be asked to sit alone in the room and tic freely for an additional 10-minutes.

SUMMARY:
Tourette syndrome (TS) is a disabling neurodevelopmental disorder characterized by motor and phonic tics. The studies proposed in this application will explore the endocrine mechanisms underlying two of the least well-understood biological characteristics of TS, namely its marked male predominance and stress susceptibility. In particular, our exploratory studies will characterize the steroid profile in TS-affected boys and girls to identify novel potential biomarkers and therapeutic targets for this disorder.

DETAILED DESCRIPTION:
Tourette syndrome (TS) is a disabling neurodevelopmental disorder characterized by motor and phonic tics. Available treatment strategies remain unsatisfactory, due to limited knowledge of the biological foundations of this disorder. The studies proposed in this application will explore the mechanisms underlying two of the least well-understood biological characteristics of TS, namely its marked male predominance and stress susceptibility. Studies from the investigators suggest that these features of TS are contributed by neuroactive steroids, a family of mediators implicated in sex and stress regulation.

The typical age of onset of TS is 6-7 years, coinciding with adrenarche, a phase of adrenal maturation characterized by an upsurge in adrenal neuroactive steroids, such as dehydroepiandrosterone (DHEA) and its sulfate (DHEAS). In preliminary studies, the investigators found that DHEA exacerbated tic-like responses in animal models of TS. Interestingly, the dose of DHEA needed to elicit TS-like responses in females is higher than those needed in males, possibly pointing to a mechanism of sex differences in TS.

Stress reduces the ability of TS patients to suppress tics, but the underlying mechanisms remain unknown. Studies in animal models indicate that this process may be due to the elevation of the neuroactive steroid allopregnanolone (AP) in the prefrontal cortex. By inhibiting the ability of the prefrontal cortex to suppress tics, AP promotes tic execution. In a pilot study, the investigators found that tic suppression, a well-known stressful task in TS patients, increases AP salivary levels. Furthermore, in another proof-of-concept study, the investigators found that inhibiting AP synthesis led to a reduction in tic severity and facilitated voluntary control of tics in stressful situations.

These findings lead to the hypothesis that TS patients exhibit alterations of the composition of their neuroactive steroid profiles, including: 1) an increase in baseline DHEA(S) levels in male TS patients, in correlation with life-time severity; and 2) an exaggerated elevation in AP in response to acute stress.

The two Aims of this proposal will test this hypothesis by: 1) comparing the baseline urinary steroidomic profile of TS-affected boys and girls with non-affected sex- and age-matched controls; and 2) charting the dynamic alterations in steroidomic salivary profiles in response to tic suppression. These studies will advance understanding of the endocrine mechanisms in TS and lead to the identification of potential biomarkers for the severity of tics and comorbid symptoms. In the long run, the results of these studies may open the way for the development of new therapies for TS that may reduce tic severity and increase patients' responsiveness to behavioral interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic criteria of TS for cases (and lack of any tic disorders for controls)
* Age between 8 and 12 years old (this age range is to ensure that TS participants can perform the tic suppression task)
* confirmation of sexual development by parent and/or self-reported Tanner stage of pubic hair development.

Exclusion Criteria:

* major psychiatric disorders such as a psychotic disorder, autism spectrum disorder, conduct disorder, and substance use disorder;
* other neurological disorders;
* clinically significant endocrinological disorders;
* use of therapies that can modify hormonal profile;
* pharmacotherapies that may change stress sensitivity, such as antidepressants and anxiolytics.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Salivary allopregnanolone concentrations | Through study completion, an average of 2 years
  Change of concentrations of salivary allopregnanolone, as measured by chromatography/ mass spectrometry. All concentrations will be expressed in pg/ml.

SECONDARY OUTCOMES:
Tic frequency | Through study completion, an average of 2 years
  Direct observation

OTHER OUTCOMES:
Measurement of salivary concentrations of other neuroactive steroids | Through study completion, an average of 2 years
  Changes in concentrations of pregnenolone, 17-hydroxypregnenolone, dehydroepiandrosterone, dehydroepiandrosterone sulfate, androstenediol, progesterone, androstenedione, testosterone, dihydroprogesterone, dihydrotestosterone, isoallopregnanolone, pregnanolone, epipregnanolone, 3-alpha androstanediol, androsterone, epiandrosterone, etiocholanolone, and cortisol as measured by chromatography/ mass spectrometry. All concentrations will be expressed in pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bortolato, MD PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No